CLINICAL TRIAL: NCT01996540
Title: The Role of Early Systematic Best Palliative Care Versus on Request Palliative Care Consultation During Standard Oncologic Treatment for Patients With Advanced Gastric or Pancreatic Cancers: a Randomized, Controlled, Multicenter Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRST100.08
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Pancreatic Neoplasm; Gastric Neoplasm
Keywords: gastric neoplasm; pancreatic neoplasm; advanced; palliative care
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional arm (Experimental): Interventional arm
  Interventions: Other: Interventional arm: Early best palliative care
- Standard arm (No Intervention): Standard arm

INTERVENTIONS:
Other: Interventional arm: Early best palliative care — Patients will receive standard oncologic care and will be assigned to early systematic best palliative care. They will meet a member of the palliative care team within 2 weeks after enrolment. Thereafter, they shall be visited by a palliative care team member every 2 weeks until death.
  Other Names: Early best palliative care
  Arms: Interventional arm

SUMMARY:
Title: The role of early systematic best palliative care versus on request palliative care consultation during standard oncologic treatment for patients with advanced gastric or pancreatic cancers: a randomized, controlled, multicenter trial.

Description of Study Treatment:

1. Interventional arm Patients will receive standard oncologic care and will be assigned to early systematic best palliative care. They will meet a member of the palliative care team within 2 weeks after enrolment. Thereafter, they shall be visited by a palliative care team member every 2 weeks until death. Patients assigned to this experimental arm will be evaluated if the total of palliative care visits between T0 (day of enrollment) and T1 (12±3 weeks) is ≥3. Palliative care visits and intervention has to be oriented by the General guidelines for palliative care: specific attention will be paid to assessing physical and psychosocial symptoms, establishing goals of care, assisting decision making regarding treatment, and coordinating care on the basis of the individual needs of the patients.

   The doctor expert in palliative care, with regular visits in the experimental arm, must be a physician dedicated full time to palliative care, that can directly prescribe drugs and other interventions, and with a particular attention to physical, psychological, and spiritual needs.

   Palliative care doctor must have the possibility to decide about organizational arrangements.

   He has to perform the palliative care visit according to Temel indications.
2. Standard arm Patients will receive standard oncologic care and will be assigned to on request palliative care consultation. They will be not scheduled to meet with the palliative care service unless a meeting will be requested by the patients, the family, or the oncologist. After the time of evaluation (T1) patients will be followed by the palliative care services as needed.

Patient completes QoL (Quality of Life) and mood questionnaires at baseline and at 12 weeks ± 3.

Patients will receive standard antineoplastic treatment in both arms of the study according to best clinical practice in each participating centre.

DETAILED DESCRIPTION:
Title: The role of early systematic best palliative care versus on request palliative care consultation during standard oncologic treatment for patients with advanced gastric or pancreatic cancers: a randomized, controlled, multicenter trial.

Short Title/Acronym: Early palliative care

Protocol Code: IRST 100.08

Study Design: randomized, controlled, multicenter trial

Study Duration: 2 years

Number of Subjects: 240

Description of Study Treatment:

1. Interventional arm Patients will receive standard oncologic care and will be assigned to early systematic best palliative care. They will meet a member of the palliative care team within 2 weeks after enrolment. Thereafter, they shall be visited by a palliative care team member every 2 weeks until death. Patients assigned to this experimental arm will be evaluated if the total of palliative care visits between T0 (day of enrollment) and T1 (12±3 weeks) is ≥3. Palliative care visits and intervention has to be oriented by the General guidelines for palliative care: specific attention will be paid to assessing physical and psychosocial symptoms, establishing goals of care, assisting decision making regarding treatment, and coordinating care on the basis of the individual needs of the patients.

   The doctor expert in palliative care, with regular visits in the experimental arm, must be a physician dedicated full time to palliative care, that can directly prescribe drugs and other interventions, and with a particular attention to physical, psychological, and spiritual needs.

   Palliative care doctor must have the possibility to decide about organizational arrangements.

   He has to perform the palliative care visit according to Temel indications.
2. Standard arm Patients will receive standard oncologic care and will be assigned to on request palliative care consultation. They will be not scheduled to meet with the palliative care service unless a meeting will be requested by the patients, the family, or the oncologist. After the time of evaluation (T1) patients will be followed by the palliative care services as needed.

Patient completes QoL (Quality of Life) and mood questionnaires at baseline and at 12 weeks ± 3.

Patients will receive standard antineoplastic treatment in both arms of the study according to best clinical practice in each participating centre.

Primary Objective:

To assess the effects on quality of life and clinical symptoms of introducing early systematic palliative care versus on request palliative care consultation during standard oncological care on quality of life.

Secondary Objectives:

* To assess the impact of early palliative care on symptom burden and mood.
* To assess the impact of families satisfaction about care.
* To compare the use of health services, including anticancer therapy, medication prescriptions, referral to hospice, hospital admissions, emergency department visits, and the location of death between study arms.
* To compare overall survival.

Statistical Methodology:

Primary endpoint is the change in the score from T0 to T1 on the Trial Outcome Index (TOI), which is the sum of the scores of specific subscale FACT-Ga or FACT-Hep concerning physical symptoms, and physical and functional well being.

Secondary endpoints are the change in the percentage of patients with anxiety and/or depression form T0 to T1 on the Mood questionnaire; the impact of families satisfaction about care; the use of health services, including anticancer therapy, medication prescriptions, referral to hospice, hospital admissions, emergency department visits, and the location of death between study arms; the overall survival.

For each type of cancer (gastric or pancreatic), we estimate that with 120 patients the study would have 80% power to detect a significant between-group difference in the change in the TOI score from T0 to T1, with a medium effect size of 0.5 standard deviation. A total of 240 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of inoperable locally advanced and/or metastatic gastric or pancreatic cancers within the previous eight weeks, any T, any N, M+ or T4 inoperable (neoadjuvant excluded);
2. patients eligible for chemotherapy and/or new target drugs treatments for metastatic or advanced disease;
3. ECOG PS 0-2 (Appendix A);
4. life expectancy >2 months;
5. both sex;
6. age ≥18 years;
7. all ethnic background;
8. subjects who are, in the opinion of the Investigator, able to understand this study and to cooperate with the study procedures;
9. written informed consent (Appendix B);
10. palliative care visit must be performed by a dedicated physician/team different from the medical oncology group.

Exclusion Criteria:

1. patients already receiving care from the palliative care service;
2. prior chemotherapy and/or new target drugs treatments for metastatic or advanced disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) | 24 months
  It is the change in the score from T0 (day of enrollment) to T1 (12±3 weeks) on the Trial Outcome Index (TOI) [which is the sum of the scores of specific subscale FACT-Ga or FACT-Hep Functional Assessment of Cancer Therapy-Gastric cancer (FACT-Ga) and Functional Assessment of Cancer Therapy-Hepatobiliary cancers (FACT-Hep) scales, concerning physical symptoms, physical and functional well being].

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 24 months
  Mood will be assessed with the use of Hospital Anxiety and Depression Scale (HADS), which is 14-item instrument composed of two subscales and screens for symptoms of anxiety and depression.
Impact of families satisfaction | 24 months
  The impact of families satisfaction about care will be evaluated by an Italian version of FAMCARE questionnaire.
Overall survival (OS) | 24 months
  It is the time from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maltoni, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (30):
- Italy (30):
  - Palliative Care Clinic IRCCS IRST, Meldola, FC
  - U.O Oncologia medica, Lugo, RA
  - S. Donato, Arezzo, Arezzo
  - Centro di Riferimento Oncologico CRO, Aviano
  - Ospedale degli Infermi,, Biella
  - Ospedale Businco, Cagliari, Cagliari
  - Policlinico Universitario, Cagliari, Cagliari
  - ASL AL, Casale Monferrato, Casale Monferrato
  - Irst-Cesena, Cesena
  - Sant'Anna, Como
  - PO M.Santo, Cosenza, Cosenza
  - Istituti Ospitalieri, Cremona, Cremona
  - Sant'Anna, Ferrara, Ferrara
  - S.Giovanni Di Dio, Firenze, Florence
  - S.Maria Annunziata,, Florence
  - E.O. Galliera, Genova
  - Aulss 12,, Mestre
  - Istituto Nazionale Tumori, Milano, Milan
  - Ospedale Sacco, Milano, Milan
  - S.PAOLO, Milan
  - IOV, Padua
  - San Matteo, Pavia
  - Guglielmo da Saliceto, Piacenza
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Fatebenefratelli,, Roma
  - SS Trinità,, Sora - Frosinone
  - Gradinego, Torino
  - AOP 9, Trapani, Trapani
  - S. Maria Gruccia, Valdarno, Valdarno
  - AULSS 12, Venezia, Venezia

REFERENCES:
- [Derived] Scarpi E, Dall'Agata M, Zagonel V, Gamucci T, Berte R, Sansoni E, Amaducci E, Broglia CM, Alquati S, Garetto F, Schiavon S, Quadrini S, Orlandi E, Casadei Gardini A, Ruscelli S, Ferrari D, Pino MS, Bortolussi R, Negri F, Stragliotto S, Narducci F, Valgiusti M, Farolfi A, Nanni O, Rossi R, Maltoni M; Early Palliative Care Italian Study Group (EPCISG). Systematic vs. on-demand early palliative care in gastric cancer patients: a randomized clinical trial assessing patient and healthcare service outcomes. Support Care Cancer. 2019 Jul;27(7):2425-2434. doi: 10.1007/s00520-018-4517-2. Epub 2018 Oct 24. PMID 30357555
- [Derived] Maltoni M, Scarpi E, Dall'Agata M, Schiavon S, Biasini C, Codeca C, Broglia CM, Sansoni E, Bortolussi R, Garetto F, Fioretto L, Cattaneo MT, Giacobino A, Luzzani M, Luchena G, Alquati S, Quadrini S, Zagonel V, Cavanna L, Ferrari D, Pedrazzoli P, Frassineti GL, Galiano A, Casadei Gardini A, Monti M, Nanni O; Early Palliative Care Italian Study Group (EPCISG). Systematic versus on-demand early palliative care: A randomised clinical trial assessing quality of care and treatment aggressiveness near the end of life. Eur J Cancer. 2016 Dec;69:110-118. doi: 10.1016/j.ejca.2016.10.004. Epub 2016 Nov 4. PMID 27821313
- [Derived] Maltoni M, Scarpi E, Dall'Agata M, Zagonel V, Berte R, Ferrari D, Broglia CM, Bortolussi R, Trentin L, Valgiusti M, Pini S, Farolfi A, Casadei Gardini A, Nanni O, Amadori D; Early Palliative Care Italian Study Group (EPCISG). Systematic versus on-demand early palliative care: results from a multicentre, randomised clinical trial. Eur J Cancer. 2016 Sep;65:61-8. doi: 10.1016/j.ejca.2016.06.007. Epub 2016 Jul 26. PMID 27472648
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/27472648 — Maltoni M et al Systematic versus on-demand early palliative care: results from a multicentre, randomised clinical trial. Eur J Cancer 2016 Sep;65:61-8
- Available data/document: study publication — https://www.ncbi.nlm.nih.gov/pubmed/27821313 — Maltoni M et al Systematic versus on-demand early palliative care: A randomised clinical trial assessing quality of care and treatment aggressiveness near the end of life. Eur J Cancer 2016 Dec;69:110-118.
- Available data/document: study publication — https://doi.org/10.1007/s00520-018-4517-2 — Scarpi E. et al Systematic vs. on-demand early palliative care in gastric cancer patients: a randomized clinical trial assessing patient and healthcare service outcomes